CLINICAL TRIAL: NCT01410955
Title: Prevention of Irinotecan Induced Diarrhea by Probiotics. A Phase III Study
Brief Title: Prevention of Irinotecan Induced Diarrhea by Probiotics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Monsea Ltd. (Industry)
Collaborators: Harmonium International Inc. (Industry); Pharma Agency (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 900450001
Record Dates: First submitted 2011-04-26; First posted 2011-08-05 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Cancer
Keywords: probiotics; diarrhoea; prevention; colon cancer; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Patients receiving probiotics.
  Interventions: Dietary Supplement: Probiotic formula
- Placebo (Placebo Comparator): Patients receiving placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic formula — Probiotic formula Colon DophilusTM , will be administered at a dose of 3x1 cps per day orally for 12 weeks. In the first cycle the starting dose is 3x1 cps per day. In other cycles the starting dose is 3x1 cps per day, or the dose according to dose adjustments from the previous treatment cycle.
  Arms: Probiotics
Dietary Supplement: Placebo — Placebo capsules will be administered at a dose of 3x1 cps per day orally for 12 weeks. In the first cycle the starting dose is 3x1 cps per day. In other cycles the starting dose is 3x1 cps per day, or the dose according to dose adjustments from the previous treatment cycle.
  Arms: Placebo

SUMMARY:
Irinotecan is one of key drug used in the treatment of colorectal cancer. The incidence of irinotecan induced diarrhea varies between 60-90%, with severe diarrhea in 20-40%. The main cause of diarrhea is one of irinotecan metabolites, SN-38 which is in the liver glucuronidated and subsequently expelled into the intestine. Due to the bacterial enzyme beta-D-glucuronidase in intestinal lumen it is deconjugated. This form causes direct damage of intestinal mucosa associated with malabsorption and the development of diarrhea. It is known that probiotic bacteria, reduce activity of intestinal beta-D-glucuronidase and therefore these bacteria could be applied in the prevention of diarrhea in patients treated by this food supplement. Given their low toxicity, good tolerability, probiotics may be an important part of supportive therapy. This is a first study aimed to determine the effectiveness of the probiotics in the prophylaxis of irinotecan induced diarrhea due to reduction intestinal beta-D-glucuronidase activity.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* histologically proven colorectal cancer patients started new line of chemotherapy based on irinotecan
* ECOG PS 0 - 1 at study entry
* life expectancy more than 3 months
* absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;

Exclusion Criteria:

* impossibility to take oral medication
* active infection treated by antibiotic therapy
* ileostomy
* hypersensitivity to study drug
* any concurrent malignancy other than non-melanoma skin cancer, no other cancer in past 5 years.
* serious concomitant systemic disorders or diseases incompatible with the study (at the discretion of investigator )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Prevention of grade 3-4 diarrhea by probiotics in patients treated by irinotecan based chemotherapy | 2 years

SECONDARY OUTCOMES:
Prevention of any grade of diarrhea | 2 years
Number of patients with any grade 3 or 4 toxicity or SAE related toxicity. | 2 years
  Number of patients with any grade 3 or 4 toxicity or SAE related toxicity according to NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE).
Number of patients with any grade gastrointestinal symptoms | 2 years
  Number of patients with any grade gastrointestinal symptoms (enteritis, colitis, constipation, abdominal distension, bloating, flatulence, gastritis, dyspepsia,nausea, vomiting) according to NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Mego, MD, PhD, Study Chair — National Cancer Institute, Slovakia; Lubos Drgona, MD, PhD, Study Chair — National Cancer Institute, Slovakia
Locations (6):
- Slovakia (6):
  - St.James Hospital and Clinic, Bardejov
  - Oncologic Institute of St.Elisabeth OUSA, Bratislava
  - National Cancer Institute, Slovakia, Bratislava
  - Zdravspol s r.o. - oncologic ambulance, Komárno
  - POKO Poprad Ltd., Poprad
  - Faculty Hospital Trencin, Trenčín